CLINICAL TRIAL: NCT02319122
Title: A Prospective Study of Two Home Based Muscle Strengthening Programs for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Svehlik Martin, MD PhD (Other)
Collaborators: University of Graz (Other)
Responsible Party: Sponsor-Investigator, Svehlik Martin, MD PhD, Senior surgeon, Medical University of Graz
Organization: Medical University of Graz (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26-526 ex 13/14
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Muscle structure; Strength training
MeSH Terms: conditions — Cerebral Palsy | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive Resistance Training (Other): The key for the PRT is the timely progression of load, based on the child's individual level of strength, which ensures progressive overload.
  Every training session will consist of a warm up, progressive resistance exercises and a cool down period. During warm up and cool down periods.These exercises will be the same for both training groups.
  The strength training exercises have been chosen to strengthen the main lower extremity muscle groups which are important for the gait: sit-to-stand, lateral step-ups, the half knee rise, heel-rises and bridging.
  All these exercises are performed loaded according to the individual level. Three sets of 8 to 10 repetitions of each exercise will be practiced on 3 non-consecutive days with moderate velocity.
  Interventions: Other: Progressive Resistance Training
- High Intensity Interval Training (Other): The High Intensity Circuit Training is a sub form of High Intensity Interval Training. The key feature is the very little rest between the exercises which causes a consistent elevation of the participant's heart rate and a short duration of the whole exercise session. Every training session consists of a warm-up, a circuit of 5 exercises (the same as these in the PRT group) and a cool-down period. The children will be asked to train 3 times a week on non-consecutive days and to perform 3 sets. Exercise workload is controlled by determination of time intervals (30 seconds). The children will be instructed to perform as many repetitions as possible during the exercise interval and to keep the rest between the exercises short (it must not exceed 30 seconds).
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — See arm description
  Other Names: HIIT
  Arms: High Intensity Interval Training
Other: Progressive Resistance Training — See arm description
  Other Names: PRT
  Arms: Progressive Resistance Training

SUMMARY:
The aim of this randomized, stratified, single-blinded study is to compare two home based strength-training protocols (High Intensity Interval Training and Progressive Resistance Training) and their effects on muscle strength, gait and aerobic and anaerobic capacity in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a common neuro-developmental disorder. Among other signs of upper motor neuron syndrome, walking pathologies and muscle weakness are leading signs of disability in children with cerebral palsy. Moreover, the gradual decline in muscle strength is part of the aging process and can be particularly devastating for people with motor disabilities. Therefore muscle-strengthening programs are indicated for children with cerebral palsy. There is evidence that lower extremity muscle strength can be increased by Progressive Resistance Training (PRT) in children with cerebral palsy. However, PRT is time consuming and therefore not always feasible for children with neurologic disorders. Moreover, it does not influence the anaerobic capacity needed for everyday activities in children. High Intensity Interval Training (HIIT) is a time efficient method, which increases both aerobic and anaerobic capacities. The aim of this randomized, stratified, single-blinded study is to compare two home based strength-training protocols (HIIT and PRT) and their effects on muscle strength, gait and aerobic and anaerobic capacity in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children with unilateral or bilateral spastic cerebral palsy
* Age between 8-16 years
* Ability to accept and follow verbal instruction
* Gross Motor Function Classification System (GMFCS) at level I-II
* Willingness to participate

Exclusion Criteria:

* Other than spastic form of cerebral palsy (ataxia, athetoid or dystonic)
* Quadriplegia
* History of orthopaedic surgery in the last 12 months
* History of Botulinum Toxin A application in the last 6 months
* Severe mental retardation

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Change in time for 6 minute Walk Test | between baseline and 2 months later (end of intervention)
  The 6 minute walk test is a self-paced, submaximal test that assesses functional capacity for walking a prolonged distance. The distance reached within 6 minutes of walking is evaluated.

SECONDARY OUTCOMES:
Change in time for Muscle Power Sprint Test | between baseline and 2 months later (end of intervention)
  Short-term muscle power will be measured using the mean power (in watts) derived from the Muscle Power Sprint Test. This test has been shown to be reliable in children with cerebral palsy. For the test, the children are instructed to complete six 15m runs at maximum pace. Between each run, the child is allowed a timed 10 second rest. Mean power output (in watts) is calculated based on the child's body weight and the average time taken to perform the six all-out sprints.
Change in Range of Motion measurements (Goniometer) | between baseline and 2 months later (end of intervention)
  Range of Motion measurements for both lower limbs.
Change in Spasticity measurements (Modified Ashworth Scale) | between baseline and 2 months later (end of intervention)
  Spasticity measurements for both lower limbs.
Change in time for Timed Up and Go Test | between baseline and 2 months later (end of intervention)
  The test requires the children to rise from an armchair stand momentarily, walk 3 meters, return to the same seat and sit down again.
Change in time for Timed Stair Test | between baseline and 2 months later (end of intervention)
  The Timed Stair Test (TST) assesses the time needed to go up and down stairs. The test is performed on a 4 or 5-step set of stairs, with handrails on both sides.
Change in Energy Expenditure Index | between baseline and 2 months later (end of intervention)
  Heart rate is an accurate and convenient measure of energy expenditure during submaximal work in normally developing children and in children with cerebral palsy and other developmental disabilities.
Change in hand held dynamometer muscle strength measurements | between baseline and 2 months later (end of intervention)
  Hand-held dynamometry (HHD) is used to quantify subjects' isometric muscle force production.
Change in Results of Dynamometry, Ultrasound imaging, Electromyography - Analysis of the muscle-tendon unit morphology and physiology measurements of the calf muscles | between baseline and 2 months later (end of intervention)
  After recording, the ultrasound images will be utilized to determine the muscle belly length, fascicle length, pennation angle and muscle thickness of the GM, muscle and tendon excursion, Achilles tendon length and cross-sectional-area (CSA) to calculate muscle and tendon stiffness and Young's modulus of the tendon.
Change in metabolomics data | between baseline and 2 months later (end of intervention)
  A metabolic profile will provide detailed information on the change in energy metabolism.
Change in results of Pediatric Outcome Data Collection Instrument (PODCI) and Activity Scale for kids performance version (ASKp) questionnaires | between baseline and 2 months later (end of intervention)
  Questionnaires measuring the childrens participation and activities of daily living (ADLs)
Change of 3D Gait Analysis data | between baseline and 2 months later (end of intervention)
  Today three dimensional segment models allow the quantification of segment and joint motions of the lower limbs in the three major planes of movement. In addition to the joint-angle and segment-position information, kinetic parameters such as joint moments and forces can be approximated.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Svehlik, MD, PhD, Principal Investigator — LKH-Univ.Klinikum Graz
Locations (1):
- LKH Graz - Department of Pediatric and Adolescent Surgery, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scholtes VA, Dallmeijer AJ, Rameckers EA, Verschuren O, Tempelaars E, Hensen M, Becher JG. Lower limb strength training in children with cerebral palsy--a randomized controlled trial protocol for functional strength training based on progressive resistance exercise principles. BMC Pediatr. 2008 Oct 8;8:41. doi: 10.1186/1471-2431-8-41. PMID 18842125
- [Background] Faigenbaum AD, Kraemer WJ, Blimkie CJ, Jeffreys I, Micheli LJ, Nitka M, Rowland TW. Youth resistance training: updated position statement paper from the national strength and conditioning association. J Strength Cond Res. 2009 Aug;23(5 Suppl):S60-79. doi: 10.1519/JSC.0b013e31819df407. PMID 19620931
- [Background] Romero-Arenas S, Martinez-Pascual M, Alcaraz PE. Impact of resistance circuit training on neuromuscular, cardiorespiratory and body composition adaptations in the elderly. Aging Dis. 2013 Oct 1;4(5):256-63. doi: 10.14336/AD.2013.0400256. PMID 24124631
- [Background] Fukumoto Y, Tateuchi H, Ikezoe T, Tsukagoshi R, Akiyama H, So K, Kuroda Y, Ichihashi N. Effects of high-velocity resistance training on muscle function, muscle properties, and physical performance in individuals with hip osteoarthritis: a randomized controlled trial. Clin Rehabil. 2014 Jan;28(1):48-58. doi: 10.1177/0269215513492161. Epub 2013 Jul 3. PMID 23823710
- [Background] Miller MB, Pearcey GE, Cahill F, McCarthy H, Stratton SB, Noftall JC, Buckle S, Basset FA, Sun G, Button DC. The effect of a short-term high-intensity circuit training program on work capacity, body composition, and blood profiles in sedentary obese men: a pilot study. Biomed Res Int. 2014;2014:191797. doi: 10.1155/2014/191797. Epub 2014 Feb 23. PMID 24707476
- [Background] Rose SA, DeLuca PA, Davis RB 3rd, Ounpuu S, Gage JR. Kinematic and kinetic evaluation of the ankle after lengthening of the gastrocnemius fascia in children with cerebral palsy. J Pediatr Orthop. 1993 Nov-Dec;13(6):727-32. doi: 10.1097/01241398-199311000-00007. PMID 8245196
- [Background] Zhao H, Ren Y, Wu YN, Liu SQ, Zhang LQ. Ultrasonic evaluations of Achilles tendon mechanical properties poststroke. J Appl Physiol (1985). 2009 Mar;106(3):843-9. doi: 10.1152/japplphysiol.91212.2008. Epub 2008 Dec 31. PMID 19118156
- [Background] Williams EN, Carroll SG, Reddihough DS, Phillips BA, Galea MP. Investigation of the timed 'up & go' test in children. Dev Med Child Neurol. 2005 Aug;47(8):518-24. doi: 10.1017/s0012162205001027. PMID 16108451
- [Derived] Schranz C, Kruse A, Tilp M, Svehlik M. Is there a relationship between muscle-tendon properties and a variety of functional tasks in children with spastic cerebral palsy? Gait Posture. 2021 Mar;85:14-19. doi: 10.1016/j.gaitpost.2021.01.009. Epub 2021 Jan 14. PMID 33487525
- [Derived] Schranz C, Kruse A, Belohlavek T, Steinwender G, Tilp M, Pieber T, Svehlik M. Does Home-Based Progressive Resistance or High-Intensity Circuit Training Improve Strength, Function, Activity or Participation in Children With Cerebral Palsy? Arch Phys Med Rehabil. 2018 Dec;99(12):2457-2464.e4. doi: 10.1016/j.apmr.2018.06.010. Epub 2018 Jul 4. PMID 30473019